CLINICAL TRIAL: NCT05138497
Title: Effects of a Program Based on High Intensity Interval Training and Low Impact on Physical, Functional, Cognitive and Psychological Condition in Colombians Older Than 65 Years.
Brief Title: HILIT on the Physical, Functional, Cognitive and Psychological Condition of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -University of Jaén
Record Dates: First submitted 2021-10-22; First posted 2021-12-01 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: For the assignment to the groups, a random sampling will be carried out from the Epidat program. This classification will be hidden, therefore, those responsible for admitting patients to the intervention phase will not know which group each has been assigned to. Said assignment will be previously carried out by a researcher who will not intervene in the subsequent phases of evaluation, data recording intervention and database development. The assignment will be communicated by sealed and totally opaque envelopes. The analysis of the results will be carried out by a researcher outside the group assignment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILIT group (Experimental): An experimental group (EG) that after an initial evaluation and with their consent, will be subjected to a directed physical training program for 12 weeks with 3 weekly sessions (Monday, Wednesday and Friday), with a duration of 50 min per session. The exercises to be carried out will be divided into three different phases: warm-up during the first 10 minutes; the main part with a duration of 30 minutes (where each exercise should be performed for 20 to 30 seconds as intense or fast as possible without generating joint impact, and then take a break for 10 to 15 seconds, before repeating it); and the return to calm, based mainly on stretching exercises with a total duration of 10 minutes.
  Interventions: Other: HILIT
- Control group (No Intervention): A control group (CG) that will not undergo treatment, which will be evaluated in the pre and post phase of the study. The participants assigned to this group will receive general advice on the positive effects of the regular practice of physical activity, and they will be given the guide of recommendations for the promotion of physical activity.

INTERVENTIONS:
Other: HILIT — A total of 92 men and women 65 years old, distributed in an experimental group that will receive a 12-week of HILIT program (n = 46); and a control group (n = 46) that will only receive general recommendations on the benefits of physical exercise. The variables will be measured for both groups with the same validated tools and the same researcher to avoid information biases and differential incorrect classification.
  Arms: HILIT group

SUMMARY:
To analyze the effects of a program based on high intensity interval training and low impact on the state of health and the physical, functional, cognitive and psychological condition in Colombian people over 65 years of age.

DETAILED DESCRIPTION:
This research corresponds to an experimental study, a double-blind randomized controlled clinical trial, where a total of 92 men and women 65 years old will be evaluated, distributed in two groups: the experimental group will receive a Beat Fit-type HILIT program (n = 46) 12 weeks; and the control group (n = 46) that will only receive general recommendations on the benefits of physical exercise. The variables will be measured for both groups with the same validated tools and the same researcher to avoid information biases and differential incorrect classification. The evaluations will be carried out at the beginning of the intervention and immediately after the end of this period, and the results will be recorded in a data record that will later be unified in an Excel database registering a code for each participant to maintain condition of privacy, but at the same time allow the required comparability.

For the independent variables, the sociodemographic characteristics, clinical history and the socio-family assessment scale will be addressed; The result variables are divided by areas: those focused on health status will measure the relative risk of death due to Comorbidity from the Charlson Index, Health-related Quality of Life [HRQoL] with the SF36 questionnaire, the Questionnaire To determine sarcopenia, it will be the SARC-F (Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls) and the Fried fragility phenotype will be applied. For the physical condition variables, the ECFA battery will be used; for the execution of sequential locomotive tasks it will be measured with the "8-foot up-and-go test"; gait and balance from the Tinetti Scale, Gait Speed with the 6-minute Test; and postural stability and balance from the Berg Scale. For the functional variables, the Katz Index (activities of daily living), the Lawton & Brody Index of the Vice-Rector's Office for Undergraduate, Postgraduate and Permanent Training (instrumental activities of daily life) and the Siu and Reuben physical scale ( Advanced activities of daily living). For the Cognitive Variable, the Minimental Status Examination (MMSE) and for the psychological variables, Yesavage will be applied for depression, the Pittsburgh Index for sleep quality and fear of falling with the international scale FES-I (Falls Efficacy Scale-International). All variables will have pre and post intervention measurements. As a result, a dance-based HILIT training program (Beat Fit) is expected to improve the health, physical, functional, cognitive and psychological condition of Colombian adults over 65 years of age, thus contributing to the comprehensive approach of this population. Once the intervention is completed, the final evaluation will be carried out and, from the comparative process, define if there are significant differences with respect to the results obtained initially.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 65 years of age, who voluntarily agree to participate in the study.
* Be able to understand the instructions and exercise protocols for this project.

Exclusion Criteria:

* Contraindications to the performance of physical tests or exercise.
* People with a diagnosis of pathologies such as cancer, pulmonary hypertension and kidney failure, a population with a diagnosis of heart failure or orphan diseases, a population with a psychiatric diagnosis and / or management, or with neurological or cognitive alterations.
* People with a diagnosis of Human Immunodeficiency Virus (HIV / AIDS) infection or disease.
* Do not agree to participate in the study or those who at the time of entry to the program have denied the endorsement of the use of their data for research in informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Charlson index. Absence of comorbidity is considered when the score is 0-1 points, low comorbidity 2 points and high cormobility in scores equal to or greater than 3 points. | Up to twelve weeks
  Relative risk of death due to comorbidity.
The Short Form-36 Health Survey (SF-36) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The results are values between 0 and 100. Optimal health is represented by scores of 100 and very poor health would equal 0.
Short Physical Performance Battery (SPPB) | Up to twelve weeks
  Short test battery, widely used in geriatrics, consists of evaluating the patient from 3 points of view: on the one hand, the patient's balance is measured, counting if he is able to maintain balance for at least 10 seconds with his feet together, in semi-tandem and tandem, counting the speed of the gait, measuring the time it takes to walk 4m, and the strength and resistance of the lower body, counting the time it takes to perform 5 squats (STS5).
The Berg Balance Scale (BBS) | Up to twelve weeks
  Used to assess a person's static and dynamic balance skills.
KATZ INDEX | Up to twelve weeks
  Is a widely used tool to assess the level of independency in older adults. It is scored considering the items grouped to obtain degrees A, B, C, etc., of independence. It is observed that 0 points are equal to grade A, 1 point to grade B, 2 points to grade C, 3 points to grade D, and so on.
  In a conventional way, the following classification can be assumed:
  * Grades A-B or 0 - 1 points = absence of disability or mild disability.
  * Grades C-D or 2 - 3 points = moderate disability.
  * Grades E-G or 4 - 6 points = severe disability.
The Lawton & Brody scale | Up to twelve weeks
  Evaluates independence and functionality in instrumental activities of daily life) such as shopping, cooking, cleaning, washing, finances, medication, transportation and use of the telephone; and considers instrumental disability the inability to perform one or more activities. Each area is scored according to the description that best corresponds to the subject. Therefore, each area scores a maximum of 1 point and a minimum of 0 points. The maximum dependence would be marked by obtaining 0 points, while a sum of 8 points would express total independence.
The physical scale of advanced life activities Reuben's day. | Up to twelve weeks
  Evaluates the degree of integration in the community, social relationships and is sensitive to the functional assessment of individuals in the community
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
MoCA (Montreal Cognitive Assessment) | Up to twelve weeks
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
The Yesavage Geriatric Depression Scale | Up to twelve weeks
  Questionnaire used to screen for depression in older people. Scores from 00 to 05 indicate Normal screening, 06 to 10 Moderate Depression screening, and 11 to 15 Severe Depression screening.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep.
FES-I (Falls Efficacy Scale-International) | Up to twelve weeks
  Questionnaire that evaluates the fear of falling. After adding the total score, values of 16-19 indicate little fear; between 20-27, intermediate fear, and from 28-64, intense fear, representing a greater risk of falls the higher the total score.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip stregth.
Tinetti scale | Up to twelve weeks
  It is used to determine early the risk of falling in an elderly person during the year following its application. The result of both sections will be added, so that a score of less than 19 points will imply a high risk of falls, a score of 19 to 24 will reflect medium risk of falls and a score of 25 to 28 will indicate low risk of falls.
TUG test (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function.

SECONDARY OUTCOMES:
SARC-F | Up to twelve weeks
  Screening to assess the risk of sarcopenia. It generates a total score of 0-10 points, of which the range of 0-3 is recorded without sarcopenia while 4-10 suggest sarcopenia.
Frailty phenotype | Up to twelve weeks
  Five original characteristics are evaluated: involuntary weight loss, self-reported exhaustion, slow gait speed, weakness, and low physical activity.
Waist circumference | Up to twelve weeks
  Is used to assess central fat distribution and degree of abdominal obesity
Hip circumference | Up to twelve weeks
  It is measured at the level of the maximum prominence of the buttocks.
Waist-to-hip ratio | Up to twelve weeks
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement
Mini Nutritional Assessment - Short Form (MNA®-SF) | Up to twelve weeks
  It is a simple and quick method to identify elderly people who are at risk of malnutrition or undernourished.
The 6-minute walk test (PC6M) | Up to twelve weeks
  Assesses in an integrated way the response of the respiratory, cardiovascular, metabolic, skeletal muscle and neurosensory systems to the stress imposed by exercise.
The 8 foot up & go test | Up to twelve weeks
  Assesses agility and dynamic balance.
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
Body Weight | Up to twelve weeks
  Is the sum of Body Fat and Fat Free Mass.
Height | Up to twelve weeks
  It measures a person's height, measured from the sole of the foot to the top of the head.

CONTACTS AND LOCATIONS:
Locations (1):
- District of agua Blanca, Santiago de Cali, Colombia